CLINICAL TRIAL: NCT02468804
Title: Cognitive Dysfunction in Parkinson's Disease
Brief Title: Cognitive Dysfunction In Parkinson's
Acronym: KL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10-0771
Record Dates: First submitted 2013-10-18; First posted 2015-06-11 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Parkinson's
Keywords: Parkinson's; Non-parkinsons
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Parkinson's Disease Subjects, (rTMS) (Experimental): The PD subjects will be randomized, and on a separate day receive a course of either real (rTMS) or sham TMS. Twenty minutes after this treatment subjects will again perform the same working memory task (at 9am to control for fatigue and diurnal effects) while having MEG data recorded
  Interventions: Device: rTMS
- Control Subjects (rTMS) (Experimental): The control subjects will be randomized, and on a separate day receive a course of either real (rTMS) or sham TMS. Twenty minutes after this treatment subjects will again perform the same working memory task (at 9am to control for fatigue and diurnal effects) while having MEG data recorded
  Interventions: Device: rTMS
- Parkinson's Disease Subjects, (sTMS) (Sham Comparator): The PD subjects will be randomized, and on a separate day receive a course of either real (rTMS) or sham TMS. Twenty minutes after this treatment subjects will again perform the same working memory task (at 9am to control for fatigue and diurnal effects) while having MEG data recorded
  Interventions: Device: Sham TMS
- Control Subjects (sTMS) (Sham Comparator): The control subjects will be randomized, and on a separate day receive a course of either real (rTMS) or sham TMS. Twenty minutes after this treatment subjects will again perform the same working memory task (at 9am to control for fatigue and diurnal effects) while having MEG data recorded
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: rTMS — TMS: Repetitive TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Stimulator (Magstim, Jali Medical US distributors, Woburn, MA). Repetitive pulses will be delivered to the right and left pre-frontal cortex (Brodman area 46) using a frameless stereotactic navigation system and the subject's MRI in Brainsight software. Stimuli will be delivered at 20 Hz at 90% of the subjects resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. The same TMS parameters as active stimulation but with the coil held at 90° to the scalp to induce similar somatic sensations and noise as in the active group with minimal direct brain effects.
  Other Names: Repetitive Transcranial Magnetic Stimulation
  Arms: Control Subjects (rTMS); Parkinson's Disease Subjects, (rTMS)
Device: Sham TMS — Sham TMS will be administered with a Magstim sham coil with electrodes attached to mimic the sounds and sensation of real TMS. The site and frequency of stimulation will be identical to the real TMS described above.
  Arms: Control Subjects (sTMS); Parkinson's Disease Subjects, (sTMS)

SUMMARY:
We hypothesize that reductions in gamma activity are a key mechanism underlying cognitive dysfunction in PD and that interventions to increase gamma activity will improve cognition.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative illness (after Alzheimer's disease) affecting 1-2% of people over age 65.3 Although PD is traditionally characterized by its motor symptoms (e.g. tremor, stiffness, slowness), research demonstrates that cognitive dysfunction has a greater impact on patient suffering and caregiver burden despite being under-recognized. Cognitive dysfunction is a significant risk factor for psychosis, dementia, nursing home placement and affects 20- 40% of PD patients even at the time of initial diagnosis.4,5 In patients with PD surviving 20 years or longer, cognitive dysfunction is the leading cause of nursing home placement and three fourths of PD patients ultimately develop dementia.6

We know that neurons in the brain communicate with each other by firing at certain frequencies. A growing literature shows that high frequency (30-50 Hz) brain activity called gamma activity is particularly important for communication between distant brain areas and is critical to normal cognition.7 Prior studies also show that gamma activity is reduced in PD.8 However, we do not know why gamma activity is reduced in PD or the relationship between changes in gamma activity and cognitive dysfunction. We hypothesize that reductions in gamma activity are a key mechanism underlying cognitive dysfunction in PD and that interventions to increase gamma activity will improve cognition.

To test this hypothesis we propose to use a novel combination of research methods including magnetoencephalography (MEG) and repetitive transcranial magnetic stimulation (rTMS). MEG measures magnetic activity over the scalp to determine brain activity. We will use MEG to determine whether reductions in gamma activity are related to cognitive dysfunction in PD. TMS uses a magnetic coil placed over the scalp to stimulate brain activity. While there is evidence that repetitive TMS (transcranial magnetic stimulation) increases gamma activity and may improve cognition, it has not been studied for this purpose in PD. We will apply repetitive TMS to PD patients to determine whether gamma activity and/or cognitive function may be improved non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit 60 PD patients through the University Colorado Hospital (UCH) Movement Disorders Clinic diagnosed with probable PD using United Kingdom (UK) Brain Bank Criteria.
* PD patients will be of mild to moderate severity based on the Hohn and Yahr scale (score of 3 or less in on medication state) and be on a stable dose of PD medications.
* Clinical severity will also be assessed using the Unified Parkinson Disease Rating Scale.
* We do not anticipate recruitment to be difficult as UCH Movement clinics see over 800 PD patients annually, the majority of whom are stage 3 or less.
* Controls will be approximately matched for age and gender as a group and recruited through clinic (spouses) and advertisements in the community.

Exclusion Criteria:

* Subjects will be excluded if they have significant depression (Beck Depression Inventory33 > 14)
* Dementia (Mini Mental State Examination34 < 26 or Frontal Assessment Battery35 < 14)
* Other neurological or psychiatric illness
* Significant history of head injury, significant systemic medical diseases (e.g. liver failure, kidney failure, poorly controlled diabetes)
* Deep Brain Stimulation (DBS)
* Cognitive enhancing medications (e.g. stimulants or acetylcholinesterase inhibitors) or contraindications to either TMS or MRI (pregnancy, pacemaker, unstable cardiac disease, skull lesion, claustrophobia, history of epilepsy or on medications known to lower seizure threshold).

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benzi Kluger, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UC Denver Building 534, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
In Progress

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI withdrawal of subjects during MEG screening:
  Several participants have ferromagnetic compounds on their body, that they cannot remove (dental work, pins or screws in bones...) but cause artifacts in the data, which prevents proper data analysis. Participants are quickly screened for artifacts during their baseline visit and possibly withdrawn.
Groups:
- Parkinson's Disease Subjects: Participants performed a working memory task during MEG recording. Then PD subjects were randomized to receive a course of either real (rTMS) or sham TMS on a separate day (max 1 week after first MEG). 20 min after TMS subjects again performed the same working memory task while having MEG data recorded
  REAL: Repetitive TMS was delivered at 20 Hz at 90% of the subjects resting motor threshold (RMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere.
  SHAM: stimulation was delivered with the same TMS parameters as active simulation but the coil held at 90 degree to the scalp to induce similar somatic sensations and noise as in the active group with minimal brain effects.
- Control Subjects: Participants performed a working memory task during MEG recording. Then control subjects were randomized to receive a course of either real (rTMS) or sham TMS on a separate day (max 1 week after first MEG). 20 min after TMS subjects again performed the same working memory task while having MEG data recorded.
  REAL: Repetitive TMS was delivered at 20 Hz at 90% of the subjects resting motor threshold (RMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere.
  SHAM: stimulation was delivered with the same TMS parameters as active simulation but the coil held at 90 degree to the scalp to induce similar somatic sensations and noise as in the active group with minimal brain effects.
Period: Overall Study
Arm/Group | Parkinson's Disease Subjects | Control Subjects
Started | 37 | 58
Completed | 36 | 50
Not Completed | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Control Subjects: Participants performed a working memory task during MEG recording. Then control subjects were randomized to receive a course of either real (rTMS) or sham TMS on a separate day (max 1 week after first MEG). 20 min after TMS subjects again performed the same working memory task while having MEG data recorded
  REAL: Repetitive TMS was delivered at 20 Hz at 90% of the subjects resting motor threshold (RMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere.
  SHAM: stimulation was delivered with the same TMS parameters as active simulation but the coil held at 90 degree to the scalp to induce similar somatic sensations and noise as in the active group with minimal brain effects.
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease Subjects | Control Subjects | Total
Number analyzed (Participants) | 36 | 50 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 45 | 70
  >=65 years | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.6) | 37 (18.1) | 47 (19.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 23 | 34
  Male | 25 | 27 | 52
Region of Enrollment [Number; unit: participants]
  United States | 36 | 50 | 86

OUTCOME MEASURES:

1. Primary Outcome: Differences in Error Rates on the NBack Task Between Real and Sham Stimulation Trials
Description: The primary cognitive outcome will be the error rates on the N-back task measured before and after real or sham TMS as a measure of working memory.
  A negative number indicates that error rate was higher (working memory skills were worse) in the sham than the real condition.
  A positive number indicates lower error rates (better working memory skills) in the sham vs real stimulation.
Time Frame: Change immediately after a single session TMS (pre will be done 1 week prior)
Measure: Mean (Standard Deviation); unit: incorrect responses
Arm/Group | Parkinson's Disease Subjects | Control Subjects
Number analyzed (Participants) | 32 | 20
incorrect responses | -0.79 (0.94) | -0.1 (1.31)

ADVERSE EVENTS:
Arm/Group | Parkinson's Disease Subjects | Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/50
Other Adverse Events (participants affected / at risk) | 1/36 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson's Disease Subjects (N=36) | Control Subjects (N=50)
headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes